CLINICAL TRIAL: NCT06572995
Title: Assessment of Intra-thoracic Water by Bio Reactance During Stabilization and Therapeutic De-escalation in Septic Shock: A Prospective, Multicenter, Observational Study
Brief Title: Thoracic Fluid Content During Stabilization and Therapeutic De-escalation in Septic Shock
Acronym: TFC-SEPSIS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC22.0275_TFC-SEPSIS
Record Dates: First submitted 2023-04-24; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Sepsis; Septic Shock; Hemodynamic Instability; Fluid Overload
MeSH Terms: conditions — Sepsis; Shock, Septic; Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In ICU, fluid challenge represents one of the cornerstones of hemodynamic care. However, fluid overload due to an excessive and/or inappropriate fluid administration could be associated with morbidity or mortality. Unfortunately, there is currently no continuous non-invasive devices to monitor fluid content at bedside. Bio reactance is a non-invasive, rapid and continuous technology developed in order to measure body fluid compartment. Monitoring devices functioning with such technology are promising to evaluate fluid overload in ICU.

DETAILED DESCRIPTION:
During the resuscitation phase of shock, fluid administration represents one of the cornerstones of care in order to increase cardiac output and improve microvascular blood flow. However, inappropriate fluid administration can increase tissue edema which compromises recovery after the resolution of shock state. Recently, Sakr et al. demonstrated that a higher fluid balance at 72 hours was associated with hospital mortality after septic shock. Furthermore, an administration of more than 5 liters of fluid during the first ICU stay was independently associated with an increase in mortality and hospital costs. Therefore, treating fluid removal appears to be a key component of the de-escalation phase of shock. Thus, all valuable parameters which potentially reflect tissue edema may help clinicians to individualized the necessity of fluid removal during the stabilization and de-escalation phase of shock. Among them, extra-vascular lung water (EVLW) measured with trans-pulmonary thermodilution is able to detect changes in thoracic fluid content but needs to be monitored invasively and only sequential values are recorded (each thermodilution measure). On the other hand, lung ultrasonography may help clinicians to assess fluid overload but its ability to quantify thoracic fluid content is difficult and subjective.

Bio reactance is a non-invasive, rapid and continuous method to measure body fluid compartment. All measures can be performed at bedside. Bio reactance monitoring devices allow measurement of hemodynamic parameters such as cardiac index or stroke volume but also Thoracic Fluid Content (TFC). TFC is measured through the changes in impedance of thoracic tissue to the electrical current. This parameter represents the whole fluid content in the thorax (intravascular, extravascular and intra-pleural). TFC has already been evaluated in several context. During hemodialysis, TFC is correlated to the amount of fluid removal and might help clinician to improve hemodialysis session management in ICU. In cardiac surgery, electrical impedance is correlated with changes in fluid balance. In ICU, TFC is able to predict a mechanical ventilation weaning failure with a moderate accuracy (AUC 0.69 [0.57 - 0.8], bet cut-off value > 50 k.Ω-1) in patients with moderate to severe alteration of left ventricular ejection fraction.

The main objective of the current study will evaluated correlation between thoracic fluid content (TFC) measurement and other valuable indices of fluid overload used at bedside. Secondary objectives will be to evaluate association between TFC and other clinical outcomes (organ dysfunction, mortality and quality of life after hospital living).

ELIGIBILITY:
Inclusion Criteria:

* Adult (Age >18 years old)
* Septic shock according to Sepsis-3 definition:

  * A suspected or confirmed infection
  * Persisting hypotension, despite adequate fluid resuscitation, requiring vasopressor to maintain a Mean Arterial Pressure (MAP) ≥ 65 mmHg
  * Lactate level > 2 mmol/l
* Predictive ICU length of stay > 3 days

Exclusion Criteria:

* Admission in ICU for more than 3 days
* Refusal to participate
* Moribund patients
* Decision of therapeutic withdrawal
* Curators

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted in ICU for septic shock
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Changes in daily body weight | Daily, during the first 10 days
  Evaluation of correlation between daily body weight and thoracic fluid content
Changes in extra vascular lung water | Daily, during the first 10 days
  Evaluation of correlation between extra vascular lung water and thoracic fluid content
Changes in daily fluid balance | Daily, during the first 10 days
  Evaluation of correlation between fluid balance and thoracic fluid content

SECONDARY OUTCOMES:
Length of ICU stay | during ICU stay (up to 10 days)
  Number of day from admission to ICU leaving
Length of hospital stay | during hospital stay (up to 10 days)
  Number of day from admission to hospital leaving
Ventilator free days at Day 28 | Day 28
  Number of day alive without mechanical from ICU admission to Day 28
Mortality at Day 28 | Day 28
  Survival (Yes/No)
Short Form-12 | 3 months
  Quality of life will measured by Short-Form 12 questionnaire. This validated scale contains sub-scale which explore eight domains: physical activities, social activities, usual role in activities, pain, mental health, emotional problem, vitality, general health perceptions. A higher Short Form-12 score is associated with a better quality of life, a lower Short Form-12 score is associated with a lower quality of life. The minimum score is 10 and the maximum is 60.
Percentage of patients who return at home | 3 months
  Evaluation of rehabilitation with the proportion of patients able to return at home
Percentage of patients who have professional activities | 3 months
  Evaluation of rehabilitation with the proportion of patients able to return at professional activities

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Chapalain, MD, Principal Investigator — University Hospital, Brest
Locations (2):
- France (2):
  - Chu Brest, Brest
  - Hegp - Aphp, Paris

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest University Hospital. Requestors will be required to sign and complete a data access agreement

REFERENCES:
- [Result] Vincent JL, De Backer D. Circulatory shock. N Engl J Med. 2013 Oct 31;369(18):1726-34. doi: 10.1056/NEJMra1208943. No abstract available. PMID 24171518
- [Result] Rivers E, Nguyen B, Havstad S, Ressler J, Muzzin A, Knoblich B, Peterson E, Tomlanovich M; Early Goal-Directed Therapy Collaborative Group. Early goal-directed therapy in the treatment of severe sepsis and septic shock. N Engl J Med. 2001 Nov 8;345(19):1368-77. doi: 10.1056/NEJMoa010307. PMID 11794169
- [Result] Marik PE, Linde-Zwirble WT, Bittner EA, Sahatjian J, Hansell D. Fluid administration in severe sepsis and septic shock, patterns and outcomes: an analysis of a large national database. Intensive Care Med. 2017 May;43(5):625-632. doi: 10.1007/s00134-016-4675-y. Epub 2017 Jan 27. PMID 28130687
- [Result] Sakr Y, Rubatto Birri PN, Kotfis K, Nanchal R, Shah B, Kluge S, Schroeder ME, Marshall JC, Vincent JL; Intensive Care Over Nations Investigators. Higher Fluid Balance Increases the Risk of Death From Sepsis: Results From a Large International Audit. Crit Care Med. 2017 Mar;45(3):386-394. doi: 10.1097/CCM.0000000000002189. PMID 27922878
- [Result] Vincent JL, Sakr Y, Sprung CL, Ranieri VM, Reinhart K, Gerlach H, Moreno R, Carlet J, Le Gall JR, Payen D; Sepsis Occurrence in Acutely Ill Patients Investigators. Sepsis in European intensive care units: results of the SOAP study. Crit Care Med. 2006 Feb;34(2):344-53. doi: 10.1097/01.ccm.0000194725.48928.3a. PMID 16424713
- [Result] Payen D, de Pont AC, Sakr Y, Spies C, Reinhart K, Vincent JL; Sepsis Occurrence in Acutely Ill Patients (SOAP) Investigators. A positive fluid balance is associated with a worse outcome in patients with acute renal failure. Crit Care. 2008;12(3):R74. doi: 10.1186/cc6916. Epub 2008 Jun 4. PMID 18533029
- [Result] Vaara ST, Korhonen AM, Kaukonen KM, Nisula S, Inkinen O, Hoppu S, Laurila JJ, Mildh L, Reinikainen M, Lund V, Parviainen I, Pettila V; FINNAKI Study Group. Fluid overload is associated with an increased risk for 90-day mortality in critically ill patients with renal replacement therapy: data from the prospective FINNAKI study. Crit Care. 2012 Oct 17;16(5):R197. doi: 10.1186/cc11682. PMID 23075459
- [Result] Jozwiak M, Silva S, Persichini R, Anguel N, Osman D, Richard C, Teboul JL, Monnet X. Extravascular lung water is an independent prognostic factor in patients with acute respiratory distress syndrome. Crit Care Med. 2013 Feb;41(2):472-80. doi: 10.1097/CCM.0b013e31826ab377. PMID 23263578
- [Result] Sakka SG, Klein M, Reinhart K, Meier-Hellmann A. Prognostic value of extravascular lung water in critically ill patients. Chest. 2002 Dec;122(6):2080-6. doi: 10.1378/chest.122.6.2080. PMID 12475851
- [Result] Bouhemad B, Zhang M, Lu Q, Rouby JJ. Clinical review: Bedside lung ultrasound in critical care practice. Crit Care. 2007;11(1):205. doi: 10.1186/cc5668. PMID 17316468
- [Result] Malbrain ML, Huygh J, Dabrowski W, De Waele JJ, Staelens A, Wauters J. The use of bio-electrical impedance analysis (BIA) to guide fluid management, resuscitation and deresuscitation in critically ill patients: a bench-to-bedside review. Anaesthesiol Intensive Ther. 2014 Nov-Dec;46(5):381-91. doi: 10.5603/AIT.2014.0061. PMID 25432557
- [Result] Kossari N, Hufnagel G, Squara P. Bioreactance: a new tool for cardiac output and thoracic fluid content monitoring during hemodialysis. Hemodial Int. 2009 Oct;13(4):512-7. doi: 10.1111/j.1542-4758.2009.00386.x. Epub 2009 Sep 16. PMID 19758300
- [Result] Perko MJ, Jarnvig IL, Hojgaard-Rasmussen N, Eliasen K, Arendrup H. Electric impedance for evaluation of body fluid balance in cardiac surgical patients. J Cardiothorac Vasc Anesth. 2001 Feb;15(1):44-8. doi: 10.1053/jcan.2001.20272. PMID 11254839
- [Result] Fathy S, Hasanin AM, Raafat M, Mostafa MMA, Fetouh AM, Elsayed M, Badr EM, Kamal HM, Fouad AZ. Thoracic fluid content: a novel parameter for predicting failed weaning from mechanical ventilation. J Intensive Care. 2020 Mar 5;8:20. doi: 10.1186/s40560-020-00439-2. eCollection 2020. PMID 32161651